CLINICAL TRIAL: NCT01173406
Title: The Efficacy of a Brief Motivational Enhancement Education Programme on Continuous Positive Airway Pressure Adherence in Obstructive Sleep Apnea: A Randomised Controlled Trial
Brief Title: Education Programme on Continuous Positive Airway Pressure Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai Yuen Kwan Agnes, Senior Technical Officer, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKCTC-1113
Record Dates: First submitted 2010-07-27; First posted 2010-08-02 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure treatment; Adherence; Education
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (SC) (Sham Comparator): Standard care
  Interventions: Behavioral: CPAP education
- Extended education (ME+SC) (Active Comparator): Motivational enhancement education + Standard care
  Interventions: Behavioral: CPAP education

INTERVENTIONS:
Behavioral: CPAP education — Standard CPAP education plus an session and one telephone follow up

SUMMARY:
The purpose of this study is to examine whether an education programme would enhance continuous positive airway pressure (CPAP) adherence.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a common sleep disorders associated with excessive daytime sleepiness and cardiovascular disease. It is prevalent both in populations of western and eastern countries. Continuous positive airway pressure (CPAP) therapy is an effective standard treatment and is widely prescribed for patients with OSA. However, the use of CPAP for such patients is disappointingly low. Low patient CPAP adherence limits the effectiveness of treatment. To determine whether there is a need for an extended education programme for the OSA patient in order to improve CPAP usage.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over.
2. Newly diagnosed of OSA and will be starting CPAP therapy

Exclusion Criteria:

1. Not suitable for CPAP therapy
2. Previously received CPAP therapy
3. Possesses restrictive and obstructive pulmonary diseases
4. Possesses hypoventilation
5. Under unstable health conditions
6. pregnant
7. History of psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
CPAP usage | 12-week
  To examine the efficacy of an education programme in enhancing the adherence of using CPAP.

SECONDARY OUTCOMES:
Daytime Sleepiness | 12-week
  To examine the efficacy of an education programme in enhancing the improvement in OSA-related health outcomes

OTHER OUTCOMES:
Self-efficacy measure for Sleep Apnea | 12-week
  To examine the efficacy of an education programe in enhancing improvement in adherence-related cognitions

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, MSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong Island, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lai AYK, Fong DYT, Lam JCM, Weaver TE, Ip MSM. The efficacy of a brief motivational enhancement education program on CPAP adherence in OSA: a randomized controlled trial. Chest. 2014 Sep;146(3):600-610. doi: 10.1378/chest.13-2228. PMID 24810282
- [Derived] Lai AY, Fong DY, Lam JC, Weaver TE, Ip MS. Linguistic and psychometric validation of the Chinese version of the self-efficacy measures for sleep apnea questionnaire. Sleep Med. 2013 Nov;14(11):1192-8. doi: 10.1016/j.sleep.2013.04.023. Epub 2013 Sep 16. PMID 24051110